CLINICAL TRIAL: NCT05233488
Title: Effect of Non-thermal Parameters of Ultrasound on Median Motor Nerve Conduction Velocity.
Brief Title: Effect of Different Ultrasound Doses on Median Nerve Conduction Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Saadeldeen Shalaby, Lecturer, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-43/02/008
Record Dates: First submitted 2022-01-29; First posted 2022-02-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Entrapment Neuropathies
Keywords: Pulsed Ultrasound; Nerve conduction parameters.
MeSH Terms: conditions — Nerve Compression Syndromes

STUDY DESIGN:
Intervention Model Description: Four groups; First group receives pulsed US 1 W/cm2 10% duty cycle. Second group receives pulsed US 1 W/cm2 50% duty cycle. Third group receives pulsed US 3 W/cm2 10% duty cycle. Fourth group receives pulsed US 3 W/cm2 50% duty cycle.
Who Masked: Participant, Care Provider
Masking Description: Participant applicator are blinded to the US dose used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low US dose (Experimental): Pulsed US, 1 W/cm2, 10% duty cycle.
  Interventions: Device: Pulsed Ultrasound Therapy
- Intermediate US dose (Experimental): Pulsed US, 1 W/cm2, 50% duty cycle.
  Interventions: Device: Pulsed Ultrasound Therapy
- High US dose (Experimental): Pulsed US, 3 W/cm2, 10% duty cycle.
  Interventions: Device: Pulsed Ultrasound Therapy
- Higher US dose (Experimental): Pulsed US, 3 W/cm2, 50% duty cycle.
  Interventions: Device: Pulsed Ultrasound Therapy

INTERVENTIONS:
Device: Pulsed Ultrasound Therapy — Ultrasound therapy is applied in the pulsed mode.

SUMMARY:
The current study investigates the effect of different doses of pulses ultrasound therapy on different nerve conduction parameters of the median nerve in healthy volunteering subjects.

DETAILED DESCRIPTION:
In the current study, we apply pulsed ultrasound therapy on median nerves of healthy volunteer subjects, at 1 W/cm2 10% duty cycle, 3 W/cm2 10% duty cycle, 1 W/cm2 50% duty cycle, and 3 w/cm2 50% duty cycle. Parameters of median nerve conduction study, Latency, amplitude, area, duration and forearm NCV are recorded before and after application of ultrasound therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 120 hands of 60 subjects of both genders with age range 18: 24 years.
2. Subjects assigned will be apparently healthy subjects with no neurological or neuromuscular history affecting the upper limb.

Exclusion Criteria:

1. Peripheral polyneuropathy.
2. Diabetes mellitus.
3. Previous surgeries or median and/or ulnar nerve release.
4. Cervical radiculopathy.
5. Median or ulnar entrapment neuropathies.
6. Previous or current pregnancies.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
CMAP distal latency | Immediately after application
  msecond
CMAP amplitude | Immediately after application
  mV
CMAP duration | Immediately after application
  msecond
Nerve conduction study | Immediately after application
  m/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Amr S Shalaby, Ph.D., Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, CSR
Time Frame: Within six months of termination of the current study.
Access Criteria: IPD sharing will be done after publication of the study results